CLINICAL TRIAL: NCT05138328
Title: Laser Treatment of Basal Cell Carcinoma Under Imaging Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David M. Ozog, Chair, Department of Dermatology, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14488
Record Dates: First submitted 2021-11-17; First posted 2021-11-30 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Carcinoma, Basal Cell
Keywords: Optical coherence tomography, reflectance confocal microscopy
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment of basal cell carcinoma with Nd:YAG laser (Experimental): All enrolled patients will be treated with the Nd:YAG laser for this study as part of the intentional intervention for this study.
  Interventions: Device: Treatment of basal cell carcinoma with Nd:YAG laser under imaging guidance of optical coherence tomography (OCT)

INTERVENTIONS:
Device: Treatment of basal cell carcinoma with Nd:YAG laser under imaging guidance of optical coherence tomography (OCT) — This will use optical coherence tomography (OCT) to assess the margins of basal cell carcinoma. Treatment will be completed by Nd:YAG laser.

SUMMARY:
This pilot study will examine the treatment of basal cell carcinoma (BCC) with laser technology under the guidance of imaging modalities to assist with surgical excision, including optical coherence tomography imaging (OCT) and reflectance confocal microscopy (RCM). The laser modality that we plan to use is the long-pulse Nd:YAG 1064nm laser, which is a nonablative laser already shown to effectively treat BCC. The addition of OCT and RCM has the opportunity to enhance outcomes by better targeting the treatment and permitting more precise monitoring of clearance. OCT is being used to enhance the effectiveness of Mohs Micrographic Surgery of these cancers by elucidating more definitive tumor margins. RCM has been shown to detect changes in the composition of cells consistent with BCC.

We propose to use these imaging devices to guide the laser treatment to achieve optimal efficacy with minimized side-effects. Primary outcome measured include complete clearance of the BCC lesion, which will be determined through clinical examination, dermoscopy, imaging (OCT and/or RCM), and saucerization biopsy. Secondary outcome variables include the significance of lesion depth (by OCT and/or RCM), lateral extent (by OCT and/or RCM), BCC type, and anatomical region on rate of clearance and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* At least one (1) biopsy-proven superficial or nodular BCC, less than or equal to 2.0 cm in largest dimension
* Willing to have photographs taken of the treatment area
* Ability to understand and carry out subject instructions or be represented by a legally authorized guardian or representative

Exclusion Criteria:

* Pregnancy
* Patients with a BCC lesion that requires excision. This would include relatively large lesions (greater than or equal to >2.0 cm diameter), lesions that penetrate deep into the skin beyond the depth of the OCT image capture, high risk lesions as defined by the American Academy of Dermatology as recurrent and sclerosing subtype BCC, or metastases.
* Subjects unable to follow-up for the full 12 months
* Subjects not willing to have biopsy taken from the treatment area
* Subjects with herpes simplex virus infection in treatment areas.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-06-12 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Clearance by imaging | 3-15 months after treatment
  Clearance of BCC as indicated by imaging of optical coherence tomography (OCT)
Clearance by biopsy | 3-15 months after treatment
  Clearance of BCC as indicated by biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No